CLINICAL TRIAL: NCT02752126
Title: A Randomized Phase III Study of Palliative Radiation of Advanced Central Tumors With Intentional Avoidance of the Esophagus
Acronym: PROACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Alexander Louie, Radiation Oncologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROACTIVE
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Esophageal sparing; Conventional radiotherapy; Palliative radiation; Central lung tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Palliative Radiation (Active Comparator): Patients in the standard arm will receive a conventional radiotherapy dose will be either 30 gray (Gy) in 10 fraction or 20Gy in 5 fractions. Patients will be stratified by intended dose prior to randomization. Radiation for patients in the standard arm should adhere to the principles of palliative radiation, with goals of alleviating symptoms or preventing potential complications.
  Interventions: Radiation: Conventional radiotherapy
- Esophageal Sparing IMRT (Experimental): Patients on the experimental arm will receive esophageal-sparing intensity-modulated radiotherapy, with the same dose(s) as in the standard arm.
  Interventions: Radiation: Esophageal-Sparing Intensity-Modulated Radiotherapy

INTERVENTIONS:
Radiation: Conventional radiotherapy — Patients will receive standard palliative radiation in dose of 30Gy in 10 fractions, or 20Gy in 5 fractions.
  Arms: Standard Palliative Radiation
Radiation: Esophageal-Sparing Intensity-Modulated Radiotherapy — Patients will receive esophageal-sparing intensity-modulated radiotherapy, of 30Gy in 10 fractions or 20Gy in 5 fractions.
  Arms: Esophageal Sparing IMRT

SUMMARY:
A randomized phase II study of palliative radiation of advanced central lung tumors with intentional avoidance of the esophagus. Patients will be randomized between standard of care palliative thoracic radiation and esophageal-sparing intensity-modulated radiation therapy (ES-IMRT) in a 1:1 ratio. Radiotherapy will be administered as soon as possible following randomization and subjects will be followed for 1 year after completion of their radiation therapy. The primary endpoint is esophageal quality of life as measured by the Esophageal Cancer Subscore (ECS) of the Functional Assessment of Cancer Therapy-Esophagus (FACT-E).

ELIGIBILITY:
Inclusion Criteria:

* American Joint Committee on Cancer (AJCC) 7th edition stage IV NSCLC or stage III not eligible for curative intent treatment
* Intended to receive palliative radiotherapy to the thorax, to a dose of 30Gy in 10 fractions or 20Gy in 5 fractions. In either treatment arm at least 5cm of the esophagus should be in the intended treatment field.
* Willingness and ability to provide informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0-3
* Age 18 years or older
* Prior or planned systemic therapy (chemotherapy, immunotherapy, targeted agents) is permissible at the discretion of the treating medical oncologist, provided that no systemic treatment is given within 2 weeks prior to RT, concurrent with RT or within a 2-week period post RT.
* Concurrent palliative RT to other metastatic sites is permissible
* Life expectancy > 3 months

Exclusion Criteria:

* Prior thoracic RT
* Serious medical comorbidities precluding RT
* Pregnant or lactating women
* Inability to attend the full course of RT or planned follow-up visits
* Planned concurrent palliative RT to the stomach and/or liver
* Congenital abnormalities of the esophagus or severe disorders of the esophagus (e.g. achalasia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06; Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Esophageal Quality of Life | 2 weeks after completion of radiotherapy
  Esophageal quality of life will be measured by the ECS of the FACT-E, measured at 2 weeks.

SECONDARY OUTCOMES:
Survival | 6 months after completion of radiotherapy
  Survival
Toxicity Rate Differences | 6 months after completion of radiotherapy
  Differences in rates of grade 2 or higher toxicity between groups will be tested using the Fisher's Exact test.
Progression-Free Survival | 6 months after completion of radiotherapy
  Differences in local/regional progression-free survival will be tested using the stratified log-rank test
Further Systemic Therapy | 6 months after completion of radiotherapy
  Differences in number of cycles of further systemic therapy will be tested using the student's t-test
Cost-Effectiveness/Utility Analysis | 6 months after completion of radiotherapy
  European Quality of Life-5 Dimensions (EQ-5D) measurements will be converted into utilities to inform cost-effectiveness/utility analysis.
Dosimetry Comparison - Gross Tumor Volume (GTV) | 6 months after completion of radiotherapy
  Dosimetric comparison of GTV will be compared using the student's t-test.
Dosimetry Comparison - Planning Target Volume (PTV) | 6 months after completion of radiotherapy
  Dosimetric comparison of PTV will be compared using the student's t-test.
Dosimetry Comparison - Pulmonary Metrics | 6 months after completion of radiotherapy
  Dosimetric comparison of standard pulmonary metrics will be compared using the student's t-test.
Dosimetry Comparison - Esophageal Metrics | 6 months after completion of radiotherapy
  Dosimetric comparison of standard esophageal metrics will be compared using the student's t-test.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - Atlantic Clinical Cancer Centre, Halifax, Nova Scotia
  - Grand River Regional Cancer Centre/Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Princess Margaret Hospital/ University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Louie AV, Granton PV, Fairchild A, Bezjak A, Gopaul D, Mulroy L, Brade A, Warner A, Debenham B, Bowes D, Kuk J, Sun A, Hoover D, Rodrigues GB, Palma DA. Palliative Radiation for Advanced Central Lung Tumors With Intentional Avoidance of the Esophagus (PROACTIVE): A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2022 Apr 1;8(4):1-7. doi: 10.1001/jamaoncol.2021.7664. PMID 35201290